CLINICAL TRIAL: NCT01199172
Title: Prospective Study of Prevention and Treatment of Voice Problems in Teachers
Brief Title: Prevention and Treatment of Voice Problems in Teachers
Acronym: Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kittie Verdolini Abbott, Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 8567; 1R01DC8567-1A2; 1R01DC008567 (NIH)
Record Dates: First submitted 2009-10-21; First posted 2010-09-10 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Voice Disorder
Keywords: Student teachers with normal or mildly disordered voices
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention)
- voice hygiene (Experimental): Subjects will receive training in voice hygiene
  Interventions: Behavioral: voice hygiene
- VH + VP (Experimental)
  Interventions: Behavioral: VH + VP

INTERVENTIONS:
Behavioral: voice hygiene — subjects will receive voice hygiene training
  Arms: voice hygiene
Behavioral: VH + VP — subjects will be trained in voice hygiene and voice production training
  Arms: VH + VP

SUMMARY:
The proposed series addresses the prevention and treatment of voice problems in teachers. Data in the literature clearly identify voice disorders as teachers' primary occupational risk not only in the U.S. but also internationally. Moreover, voice problems constitute a global women's health concern. Until recently, few reports have been available around the treatment of these problems in teachers, and even fewer have addressed the equally important question of prevention. The present studies are conducted within the context of a long-range goal to identify effective intervention methodologies for both the prevention and treatment of voice problems in teachers taking into consideration multicultural and linguistic factors. The present studies will report pragmatic data around the effectiveness of two theoretically-driven approaches to the prevention and treatment of voice problems in teachers, (a) voice hygiene education (VH) and (b) voice hygiene education + voice production training in "resonant voice" (VH+VP, essentially the Lessac-Madsen Resonant Voice Therapy program). Participants will be student teachers in Pittsburgh and Hong Kong, who will be followed from student teaching across their second full year of employment as a professional teacher. The central aims are: [1] to evaluate the effectiveness of VH and VH+VP for the prevention of future voice problems in student teachers who are vocally healthy at the outset of the protocol, versus the treatment of voice problems in student teachers who already have them at some level; [2] to evaluate the generality of the findings across teachers in the U.S. and China, using appropriate linguistic and cultural adaptations of the interventions; and [3] to evaluate the feasibility of an internet-based voice exercise and reporting program as a supplement to face-to-face interventions. Ergonomic and personal factors will also be evaluated for their differential ability to predict the risk for future voice problems in teachers. The results should be useful at a practical level, and should also lay the groundwork for future studies assessing similar issues around the prevention of voice problems in teachers, in particular as influenced by multicultural factors within the U.S. The results should also be useful for future studies investigating causal pathways in interventions around these problems.

ELIGIBILITY:
By self-report in person or over the phone: (a) 21-40 yr; (b) no current self-perceived voice problem;(c) student teacher in the final year of formal education prior to the initiation of employment as a teacher and imminent start of the first formal teaching practicum; (d) availability and willingness to attend up to an 8-hr group intervention on 1 of 2 days when it will be offered the week before the start of student teaching, willingness to be randomized to one of three groups, and stated willingness to persist with the entire 2.5-yr protocol, which will involve baseline, 1-mo, 3-mo, 1-yr,and 2-yr follow-up measures, and two separate interventions followed by a 4-wk hygiene reporting and potentially voice exercise period for intervention groups; (e) intention to obtain employment as a teacher in the school year following graduation; (f) no degenerative or other medical conditions or medications that would affect voice, with the exception of seasonal allergies (and their treatment) or laryngopharyngeal reflux (LPR; and its treatment).

· By clinical evaluation, for students satisfying the self-report criteria: (g) nasal patency sufficient at least unilaterally for the passage of a flexible scope; (h) no history or suspected allergy to any local anesthetic or evidence that a laryngeal exam can be conducted without it; (i) acceptably controllable gag reflex; (j) overall voice quality score < 15 on a 100-mm visual analogue scale, following standardized procedures (see D.2.4.1), together with a total VHI score < 17 and normal larynx (D.2.4.1; "low-starter group"-assuming the subject has indicated normal voice by self report, or overall voice quality score < 20, together with a total VHI score > 25 and either normal larynx or mildly impaired larynx not held to require clinical attention outside the auspices of the protocol(D.2.4.1; "high-starter group")-if the subject has indicated normal voice or at most mild, intermittent voice problems by self report; and (k) normal hearing bilaterally (30 dB at 125, 250, 500, 1000, 2000, 4000, and 8000 Hz in the better ear).

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2009-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Voice Handicap Index | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States